CLINICAL TRIAL: NCT05995249
Title: A Phase 1, 3-Part, Open-label, Drug-Drug Interaction Study to Evaluate the Effect of a Moderate CYP3A4 Inhibitor, and of Strong and Moderate CYP3A4 Inducers on the Pharmacokinetics of TAK-279 in Healthy Subjects
Brief Title: A Study of the Interaction of TAK-279 With Substances That Have an Impact on Metabolism in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: TAK-279-1002
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — Erythromycin; Phenytoin; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1, Treatment A + Treatment B: TAK-279 50 mg + Erythromycin 500 mg (Experimental): Participants will receive single oral dose of TAK-279 50 mg, on Day 1 of Period 1. Following Period 1 participants will receive single oral dose of TAK-279 50 mg, on Day 5 and erythromycin 500 mg orally thrice daily (TID) on Day 1 through Day 10 of Period 2 in Part 1 of the study.
  Interventions: Drug: TAK-279; Drug: Erythromycin
- Part 2, Treatment C + Treatment D: TAK-279 50 mg + Phenytoin 100 mg (Experimental): Participants will receive single oral dose of TAK-279 50 mg, on Day 1 of Period 1. Following Period 1 participants will receive single oral dose of TAK-279 50 mg on Day 14 and phenytoin 100 mg orally TID on Day 1 through Day 18 of Period 2 in Part 2 of the study.
  Interventions: Drug: TAK-279; Drug: Phenytoin
- Part 3, Treatment E + Treatment F: TAK-279 50 mg + Efavirenz 600 mg (Experimental): Participants will receive single oral dose of TAK-279 50 mg, on Day 1 of Period 1. Following Period 1 participants will receive single oral dose of TAK-279 50 mg on Day 11 and efavirenz 600 mg orally once daily (QD) on Day 1 through Day 15 of Period 2 in Part 3 of the study.
  Interventions: Drug: TAK-279; Drug: Efavirenz

INTERVENTIONS:
Drug: TAK-279 — TAK-279 capsules
Drug: Erythromycin — Erythromycin tablets
  Arms: Part 1, Treatment A + Treatment B: TAK-279 50 mg + Erythromycin 500 mg
Drug: Phenytoin — Phenytoin capsules
  Arms: Part 2, Treatment C + Treatment D: TAK-279 50 mg + Phenytoin 100 mg
Drug: Efavirenz — Efavirenz tablets
  Arms: Part 3, Treatment E + Treatment F: TAK-279 50 mg + Efavirenz 600 mg

SUMMARY:
The main aim of this study is to find out how the body of a healthy adult processes TAK-279 (pharmacokinetics) when substances that either hinder or help the human metabolism such as erythromycin, phenytoin and efavirenz are given along with TAK-279. Other aim is to learn about side effects and how well it is tolerated when TAK-279 is given alone and together with substances that impact human metabolism.

The participants will need to stay at the clinic for up to 26 days.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-279. TAK-279 is being tested to assess the effect of a moderate CYP3A4 inhibitor (erythromycin- Part 1), and of strong (phenytoin- Part 2) and moderate (efavirenz- Part 3) CYP3A4 inducers on the pharmacokinetics of TAK-279 in healthy participants.

The study will enroll approximately 48 patients. Participants will be enrolled in one of the three parts to receive a single dose of TAK-279 in both Period 1 and Period 2 along with multiple doses of either erythromycin, phenytoin or efavirenz in Period 2 as given below:

* Part 1, Treatment A + Treatment B: TAK-279 50 mg + Erythromycin 500 mg
* Part 2, Treatment C + Treatment D: TAK-279 50 mg + Phenytoin 100 mg
* Part 3, Treatment E + Treatment F: TAK-279 50 mg + Efavirenz 600 mg

All participants will be monitored for up to 14 days postdose in each Part.

This single-center trial will be conducted in the United States. The overall study duration is approximately 65 days for Part 1, 73 days for Part 2, and 70 days for Part 3.

ELIGIBILITY:
Inclusion criteria:

1. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.
2. Healthy, adult, male or female of non-childbearing potential, 18-55 years of age, inclusive, at the screening visit.
3. Male participants must follow protocol specified contraception guidance.
4. Continuous non-smoker who has not used nicotine- and tobacco-containing products for at least 3 months prior to the first dosing based on participant self-reporting.
5. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m^2 at the screening visit.
6. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, and electrocardiograms (ECGs), as deemed by the Investigator or designee, including the following:

   * Seated blood pressure (BP) is ≥ 90/40 millimeter of mercury (mmHg) and ≤ 140/90 mmHg at the screening visit.
   * Seated pulse rate is ≥ 40 beats per minute (bpm) and ≤ 99 bpm at the screening visit.
   * Part 1 only: QTcF interval is ≤ 450 msec (males and females) and has ECG findings considered normal or not clinically significant by the Investigator or designee at the screening visit.
   * Part 2 and 3: ECG findings considered normal or not clinically significant by the Investigator or designee at the screening visit.
   * Estimated glomerular filtration rate (eGFR) ≥ 80 mL/min/1.73m^2 at the screening visit.
   * Liver function tests including Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase (ALP), and total bilirubin ≤ upper limit of normal (ULN) at the screening visit and at check-in.
   * No clinically significant hypokalemia or hypomagnesemia at the screening visit.

Exclusion criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
3. History of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
4. Has a history of any of the following:

   * Active infection or febrile illness within 7 days prior to first dosing, as assessed by the Investigator or designee.
   * Symptoms suggestive of systemic or invasive infection requiring hospitalization or treatment within 8 weeks prior to first dosing.
   * Chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, or chronic skin ulcerations/infections or fungal infections (except superficial nailbed mycosis).
   * An infected joint prosthesis unless that prosthesis has been removed or replaced greater than 60 days prior to first dosing.
   * Opportunistic infections (eg, Pneumocystis jirovecii pneumonia, histoplasmosis, coccidiomycosis).
   * Cancer or lymphoproliferative disease within 5 years prior to first dosing, with the exception of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix is not exclusionary.
   * Known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency; splenectomy.
   * Liver or other solid organ transplant.
5. Has history or presence of alcoholism and/or drug abuse within the past 2 years prior to first dosing, as determined by the Investigator or designee.
6. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs, including macrolide antibiotics (Part 1 only; eg, erythromycin) or anti-seizure agents (Part 2 only; eg, phenytoin) or anti-viral drugs (Part 3 only; eg, efavirenz).
7. Part 2 and Part 3 only: Any positive responses on the Columbia-Suicide Severity Rating Scale (C-SSRS) or has a risk of suicide according to the Investigator's or designee judgment based on the assessment of the C-SSRS at the screening visit or check-in or has made a suicide attempt within 12 months before the first dosing.
8. Part 2 only: History of seizure (excluding simple febrile seizure), epilepsy, severe head injury, multiple sclerosis, or other known neurological conditions which the Investigator or designee considers to be clinically significant.
9. Part 2 only: Participant is known to be a CYP2C9 and/or CYP2C19 poor metabolizer based on genotyping prior to screening or is determined to be a CYP2C9 and/or CYP2C19 poor metabolizer at the screening visit.
10. History or presence of ventricular dysfunction or risk factors for Torsades de Pointes (eg, heart failure, cardiomyopathy, family history of Long QT Syndrome).
11. Female participant of childbearing potential.
12. Female participant with a positive pregnancy test at the screening visit or at check-in or who is lactating.
13. Positive urine drug or alcohol results at the screening visit or check-in.
14. Unable to refrain from or anticipates the use of:

    * Any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing.
    * Any drugs known to be moderate or strong inducers of CYP3A4 enzymes and/or P-glycoprotein (P-gp), including St. John's Wort, for 28 days prior to the first dosing. Appropriate sources (eg, Flockhart Table™) including the product label for erythromycin (Erythromycin Tablets USP 2018), phenytoin (DILANTIN (extended phenytoin sodium capsules) 2022), and efavirenz (SUSTIVA (efavirenz) capsules and tablets 2019) will be consulted to confirm lack of pharmacokinetic (PK)/pharmacodynamic interaction with the study drugs.
15. Has been on a diet incompatible with the on study diet, in the opinion of the Investigator or designee, within the 30 days prior to first dosing and throughout the study.
16. Has made a donation of blood or had significant blood loss within 56 days prior to first dosing.
17. Has made a plasma donation within 7 days prior to first dosing.
18. Participated in another clinical study within 30 days prior to first dosing. The 30 day window will be derived from the date of the last dosing in the previous study to Day 1 of Period 1 of the current study.
19. Herpes infections:

    * Participant has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at screening or Day 1 of Period 1.
    * Participant has history of serious herpetic infection that includes any episode of disseminated disease, multidermatomal herpes simplex virus, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
20. Positive results for non-herpetic viral diseases at the screening visit:

    * Hepatitis C virus (HCV) antibody and a positive confirmatory test result for HCV ribonucleic acid (RNA) (nucleic acid test or polymerase chain reaction [PCR]);
    * Hepatitis B surface antigen (HBsAg)+, hepatitis B virus deoxyribonucleic acid (DNA), or HBcAb+ with positive hepatitis B virus DNA;
    * Human immunodeficiency virus (HIV).
21. Positive results for tuberculosis (TB) at the screening visit or has the following:

    * Has history of active TB infection, regardless of treatment status.
    * Has signs or symptoms of active TB (including but not limited to chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the investigator or designee.
    * Has evidence of latent tuberculosis infection (LTBI) as evidenced by a positive QFT result OR 2 indeterminant Quantiferon TB Gold (QFT) results and does not have documentation of appropriate LTBI prophylaxis. Participant remains eligible if he or she can provide documentation of prior and complete treatment for LTBI (appropriate in duration and type per current local country guidelines).
    * Has had any imaging study during or 6 months prior to screening, including x-ray, chest computed tomography, magnetic resonance imaging, or other chest imaging suggesting evidence of current active or a history of active TB.
22. Part 3 only: History of amphetamine and methylphenidate use; history or presence of sleeping disorders or sleeping irregularities, or any significant cardiac abnormality in the opinion of the Investigator or designee.
23. Part 2 and Part 3 only: History or presence of Stevens-Johnson Syndrome and/or seizures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Parts 1, 2, and 3: Cmax: Maximum Observed Plasma Concentration for TAK-279 | Predose and at multiple timepoints post dose from Day 1 period 1 (length= 6 days) to period 2 Day 11 in Part 1 (length= 11 days), up to period 2 Day 19 in Part 2 (length= 19 days) and up to period 2 Day 16 in Part 3 (length= 16 days)
Parts 1, 2, and 3: AUC∞: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for TAK-279 | Predose and at multiple timepoints post dose from Day 1 period 1 (length= 6 days) to period 2 Day 11 in Part 1 (length= 11 days), up to period 2 Day 19 in Part 2 (length= 19 days) and up to period 2 Day 16 in Part 3 (length= 16 days)
Parts 1, 2, and 3: AUClast: Area Under the Plasma Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration for TAK-279 | Predose and at multiple timepoints post dose from Day 1 period 1 (length= 6 days) to period 2 Day 11 in Part 1 (length= 11 days), up to period 2 Day 19 in Part 2 (length= 19 days) and up to period 2 Day 16 in Part 3 (length= 16 days)

SECONDARY OUTCOMES:
Parts 1, 2, and 3: Number of Participants with Treatment-emergent Adverse Events (TEAEs) | From Day 1 of period 1 through period 2 Day 11 (up to approximately 65 days) in Part 1, up to period 2 Day 19 (up to approximately 73 days) in Part 2 and up to period 2 Day 16 (up to approximately 70 days) in Part 3
Parts 1, 2, and 3: Number of Participants with Abnormal Vital Signs | From Day 1 of period 1 through period 2 Day 11 (up to approximately 65 days) in Part 1, up to period 2 Day 19 (up to approximately 73 days) in Part 2 and up to period 2 Day 16 (up to approximately 70 days) in Part 3
  Abnormal vital sign assessment will include assessments of systolic and diastolic blood pressure, pulse rate, respiration rate, body temperature as determined by the investigator.
Parts 1, 2, and 3: Number of Participants with Abnormal Electrocardiogram Findings | From Day 1 of period 1 through period 2 Day 11 (up to approximately 65 days) in Part 1, up to period 2 Day 19 (up to approximately 73 days) in Part 2 and up to period 2 Day 16 (up to approximately 70 days) in Part 3
  Abnormal 12-lead ECG findings will include heart rate and measures PR, QRS, QT and QTcF intervals. 12-lead ECG recordings were obtained after the participants have rested for at least 5 minutes in supine position as determined by the investigator.
Parts 1, 2, and 3: Number of Participants with Abnormal Laboratory Values | From Day 1 of period 1 through period 2 Day 11 (up to approximately 65 days) in Part 1, up to period 2 Day 19 (up to approximately 73 days) in Part 2 and up to period 2 Day 16 (up to approximately 70 days) in Part 3
  Abnormal laboratory investigation will include hematology, chemistry, and urinalysis analysis as determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion - Tempe, AZ Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/903b04f400364845?idFilter=%5B%22TAK-279-1002%22%5D